CLINICAL TRIAL: NCT01545076
Title: Randomized, Multicenter, Double-blind, Placebo-controlled, Parallel-group Phase III Study to Investigate the Efficacy, Safety, and Tolerability of 2 Different Doses of IgPro20 (Subcutaneous Immunoglobulin) for the Treatment of Chronic Inflammatory Demyelinating Polyneuropathy (CIDP) - the PATH Study
Brief Title: Chronic Inflammatory Demyelinating Polyneuropathy (CIDP) and Treatment With Subcutaneous Immunoglobulin (IgPro20)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Collaborators: ICON Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IgPro20_3003
Record Dates: First submitted 2012-03-01; First posted 2012-03-06 (Estimated); Results first posted 2018-07-05 (Actual); Last update posted 2018-07-05 (Actual); Status verified 2016-12

CONDITIONS: Chronic Inflammatory Demyelinating Polyneuropathy; Polyradiculoneuropathy
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating; Polyradiculoneuropathy | interventions — Hizentra

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- IgPro20 low dose (Experimental)
  Interventions: Biological: IgPro20 (low dose); Biological: IgPro10
- IgPro20 high dose (Experimental)
  Interventions: Biological: IgPro10; Biological: IgPro20 (high dose)
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo; Biological: IgPro10

INTERVENTIONS:
Biological: IgPro20 (low dose) — 20% liquid formulation (200 mg/mL) of human normal immunoglobulin for subcutaneous use administered weekly during the SC treatment period of the study according to the randomization:
  0.2 g/kg body weight (low dose arm)
  Other Names: Hizentra
  Arms: IgPro20 low dose
Biological: Placebo — 2% human albumin administered by weekly SC infusions during the SC treatment period of the study.
  Arms: Placebo
Biological: IgPro10 — 10% Immunoglobulin G (IgG) liquid formulation of human normal immunoglobulin (Privigen®) administered intravenously during Restabilization Period of the study and/or as Rescue Therapy during SC Treatment Period for subjects with a CIDP relapse.
Biological: IgPro20 (high dose) — 20% liquid formulation (200 mg/mL) of human normal immunoglobulin for subcutaneous use administered weekly during the SC treatment period of the study according to the randomization:
  0.4 g/kg body weight (high dose arm)
  Other Names: Hizentra
  Arms: IgPro20 high dose

SUMMARY:
This is a prospective, multicenter, randomized, double-blind, placebo-controlled, parallel-group 3-arm study to investigate 2 different doses of subcutaneous (SC) IgPro20 compared with placebo for maintenance treatment of patients with CIDP.

Patients who received at lease 1 dose of intravenous immunoglobulin (IVIG) within 8 weeks before screening will be assessed during 4 separate study periods. Patients first undergo a Screening Period, followed by an IgG Dependency Test Period of up to 12 weeks to test for ongoing need of IgG. Those patients experiencing CIDP relapse during this test period will be administered a standardized IVIG regimen during an IVIG Re-stabilization Period. Patients with improved and maintained adjusted inflammatory neuropathy cause and treatment scale (INCAT) in the IVIG Re-stabilization Period will continue to the SC Treatment Period of the study. Patients entering the 24 week SC Treatment Period will be randomized to receive weekly infusions of 1 of 2 IgPro20 doses (0.2 or 0.4 g/kg body weight) or placebo.

The overall study duration is up to 52 weeks. Clinical outcomes will be assessed by the Inflammatory Neuropathy Cause and Treatment (INCAT) score, maximum grip strength, the Medical Research Council (MRC) sum score, the Rasch-built Overall Disability Scale (R-ODS), and electrophysiological evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Definite or probable CIDP according to the European Federation of Neurological Societies/Peripheral Nerve Society (EFNS/PNS) criteria 2010.
* An IVIG treatment during the last 8 weeks prior to enrollment.
* Age ≥18 years.
* Written informed consent for study participation obtained before undergoing any study-specific procedures.

Exclusion Criteria:

* Any polyneuropathy of other causes
* Any other disease (mainly neurological or chronic orthopedic) that has caused neurological symptoms or may interfere with treatment or outcome assessments
* Severe diseases and conditions that are likely to interfere with evaluation of the study product or satisfactory conduct of the study
* History of thrombotic episodes within the 2 years prior to enrolment
* Known allergic or other severe reactions to blood products including intolerability to previous IVIG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2012-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Ivo N. van Schaik, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (91):
- United States (22):
  - Site reference 8400181, Birmingham, Alabama
  - Site reference 8400173, Phoenix, Arizona
  - Site reference 8400172, Phoenix, Arizona
  - Site reference 8400167, Los Angeles, California
  - Site reference 8400077, Centennial, Colorado
  - Site Reference 8400352, Washington D.C., District of Columbia
  - Site reference 8400214, Miami, Florida
  - Site reference 8400162, Chicago, Illinois
  - Site Reference 8400247, Chicago, Illinois
  - Site Reference 8400215, Indianapolis, Indiana
  - Site reference 8400166, Kansas City, Kansas
  - Site Reference 8400347, New Brunswick, New Jersey
  - Site reference 8400169, New York, New York
  - Site reference 8400179, New York, New York
  - Site reference 8400182, Charlotte, North Carolina
  - Site Reference 8400346, Durham, North Carolina
  - Site reference 8400178, Columbus, Ohio
  - Site reference 8400217, Oklahoma City, Oklahoma
  - Site Reference 8400177, Nashville, Tennessee
  - Site reference 8400164, Houston, Texas
  - Site Reference 8400268, Charlottesville, Virginia
  - Site Reference 8400340, Seattle, Washington
- Australia (3):
  - Site Reference 0360017, Herston, Queensland
  - Site reference 0360011, Fitzroy, Victoria
  - Site reference 0360008, Southport
- Site reference 0560003, Leuven, Belgium
- Canada (5):
  - Site Reference 1240048, Vancouver, British Columbia
  - Site Reference 1240051, Montreal, Quebec
  - Site reference 1240006, Edmonton
  - Site reference 1240007, Québec
  - Site reference 1240009, Toronto
- Czechia (3):
  - Site reference 2030002, Hradec Králové
  - Site reference 2030009, Hradec Králové
  - Site reference 2030003, Prague
- Estonia (2):
  - Site Reference 2330002, Tallinn
  - Site Reference 2330003, Tallinn
- Site reference 2460002, Helsinki, Finland
- France (4):
  - Site reference 2500024, Clermont-Ferrand
  - Site reference 2500013, Marseille
  - Site reference 2500022, Nice
  - Site reference 2500019, Pessac
- Germany (15):
  - Site reference 2760048, Berlin
  - Site reference 2760069, Berlin
  - Site reference 2760072, Berlin
  - Site reference 2760049, Bochum
  - Site reference 2760080, Cologne
  - Site reference 2760075, Düsseldorf
  - Site Reference 2760094, Essen
  - Site reference 2760052, Essen
  - Site reference 2760036, Göttingen
  - Site reference 2760053, Göttingen
  - Site reference 2760054, Hanover
  - Site Reference 2760113, Ibbenbueren
  - Site reference 2760055, Leipzig
  - Site reference 2760047, Potsdam
  - Site reference 2760039, Würzburg
- Israel (2):
  - Site reference 3760005, Haifa
  - Site reference 3760002, Tel Aviv
- Italy (8):
  - Site reference 3800026, Chieti
  - Site reference 3800027, Florence
  - Site reference 3800028, Genova
  - Site reference 3800031, Milan
  - Site reference 3800035, Roma
  - Site reference 3800036, Roma
  - Site reference 3800030, Rozzano
  - Site reference 3800037, Torino
- Japan (12):
  - Site Reference 3920040, Aomori
  - Site Reference 3920042, Aomori
  - Site reference 3920038, Chiba
  - Site reference 3920061, Kanagawa
  - Site reference 3920045, Matsumoto
  - Site reference 3920058, Osaka
  - Site reference 3920037, Saitama
  - Site reference 3920034, Tokushima
  - Site Reference 3920065, Tokyo
  - Site Reference 3920062, Tokyo
  - Site reference 3920032, Tokyo
  - Site reference 3920035, Yamaguchi
- Netherlands (3):
  - Site reference 5280001, Amsterdam
  - Site reference 5280005, Maastricht
  - Site reference 5280004, Utrecht
- Poland (3):
  - Site Reference 6160058, Gdansk
  - Site Reference 6160060, Lodz
  - Site Reference 6160055, Lublin
- Spain (5):
  - Site reference 7240010, Barcelona
  - Site reference 7240011, Barcelona
  - Site reference 7240013, Madrid
  - Site reference 7240014, Madrid
  - Site reference 7240016, Seville
- United Kingdom (2):
  - Site reference 8260019, London
  - Site Reference 8260032, Manchester

REFERENCES:
- [Derived] van Schaik IN, Bril V, van Geloven N, Hartung HP, Lewis RA, Sobue G, Lawo JP, Praus M, Mielke O, Durn BL, Cornblath DR, Merkies ISJ; PATH study group. Subcutaneous immunoglobulin for maintenance treatment in chronic inflammatory demyelinating polyneuropathy (PATH): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Neurol. 2018 Jan;17(1):35-46. doi: 10.1016/S1474-4422(17)30378-2. Epub 2017 Nov 6. PMID 29122523
- [Derived] van Schaik IN, van Geloven N, Bril V, Hartung HP, Lewis RA, Sobue G, Lawo JP, Mielke O, Cornblath DR, Merkies IS; PATH study group. Subcutaneous immunoglobulin for maintenance treatment in chronic inflammatory demyelinating polyneuropathy (The PATH Study): study protocol for a randomized controlled trial. Trials. 2016 Jul 25;17(1):345. doi: 10.1186/s13063-016-1466-2. PMID 27455854

RESULTS

PARTICIPANT FLOW:
Groups:
- IgPro10 Re-stabilization: Subjects who experienced CIDP qualified for IVIG re-stabilization treatment with IgPro10 (10% IgG preparation for intravenous administration).
- IgPro20 (0.4): Subjects completing IVIG re-stabilization went on to the IgPro20 Subcutaneous (SC) Treatment. IgPro20 [0.4 g/kg body weight (bw)]: 20% liquid formulation (200 mg/mL) of human normal immunoglobulin for subcutaneous use administered weekly.
- IgPro20 (0.2): Subjects completing IVIG re-stabilization went on to the IgPro20 Subcutaneous (SC) Treatment. IgPro20 [0.2 g/kg body weight (bw)]: 20% liquid formulation (200 mg/mL) of human normal immunoglobulin for subcutaneous use administered weekly.
- Placebo: Subjects completing IVIG re-stabilization went on to the IgPro20 Subcutaneous (SC) Treatment. Placebo: 2% human albumin administered by weekly SC infusions.
- IgPro10 Rescue: Subjects with CIDP relapse during the SC Treatment Period received IgPro10 (10% IgG preparation for intravenous administration) as rescue medication.
Period: IgPro10 Restabilization Period
Arm/Group | IgPro10 Re-stabilization | IgPro20 (0.4) | IgPro20 (0.2) | Placebo | IgPro10 Rescue
Started | 208 | 0 | 0 | 0 | 0
Completed | 172 | 0 | 0 | 0 | 0
Not Completed | 36 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 4 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0
Not completed — Failure to meet randomization criteria | 22 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 0 | 0 | 0 | 0
Period: IgPro20 Subcutaneous Treatment Period
Arm/Group | IgPro10 Re-stabilization | IgPro20 (0.4) | IgPro20 (0.2) | Placebo | IgPro10 Rescue
Started | 0 | 58 | 57 | 57 | 0
Completed | 0 | 39 | 36 | 21 | 0
Not Completed | 0 | 19 | 21 | 36 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 10 | 18 | 32 | 0
Not completed — Adverse Event | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 8 | 2 | 3 | 0
Period: IgPro10 Rescue Period
Arm/Group | IgPro10 Re-stabilization | IgPro20 (0.4) | IgPro20 (0.2) | Placebo | IgPro10 Rescue
Started | 0 | 0 | 0 | 0 | 60
Completed | 0 | 0 | 0 | 0 | 60
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Pre-randomization Safety Data Set (PSDS): The PSDS was based on all subjects enrolled into the study who received at least 1 dose of IgPro10 (in the re-stabilization period) before randomization into the subcutaneous period. One subject withdrew from the re-stabilization period prior to receiving IgPro10, therefore n=207 for the PSDS.
Groups:
- Pre-randomization Safety Data Set (PSDS): Pre-randomization Safety Data Set (PSDS): The PSDS was based on all subjects enrolled into the study who received at least 1 dose of IgPro10 (in the re-stabilization period) before randomization into the subcutaneous period. One subject withdrew from the re-stabilization period prior to receiving IgPro10, therefore n=207 for the PSDS.
Arm/Group | Pre-randomization Safety Data Set (PSDS)
Number analyzed (Participants) | 207
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 150
  >=65 years | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (12.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76
  Male | 131
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25
  Czechia | 6
  Japan | 15
  United Kingdom | 6
  Spain | 16
  Canada | 19
  Netherlands | 7
  Belgium | 2
  Finland | 1
  Poland | 8
  Italy | 32
  Israel | 2
  Australia | 6
  France | 9
  Germany | 51
  Estonia | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage (%) of Subjects With CIDP Relapse or Are Withdrawn for Any Other Reason During the Subcutaneous (SC) Treatment Period
Description: Relapse is defined as an increase of at least 1 INCAT score point (except for the increase from 0 to 1 in the upper limb score). The INCAT score is a 10-point scale that covers the functionality of legs and arms, and has been successfully used to measure treatment effects in various CIDP studies. Scores for arm disability range from 0 ("No upper limb problems") to 5 ("Inability to use either arm for any purposeful movement"), and scores for leg disability range from 0 ("Walking not affected") to 5 ("Restricted to wheelchair, unable to stand and walk a few steps with help"). The INCAT (total) score is the sum of these 2 scores and ranges from 0 to 10. For the "adjusted" INCAT score, changes in the function of the upper limbs from 0 (normal) to 1 (minor symptoms) or from 1 to 0 were not recorded as deterioration or improvement because these changes are not considered clinically significant.
Time Frame: Up to 25 weeks
Population: Intention-to-treat Set (ITTS): The ITTS consists of all randomized subjects who received at least 1 dose of IgPro20 / placebo and satisfied inclusion criterion #1 (diagnosis of CIDP).
Measure: Number; unit: percentage of subjects
Groups:
- IgPro20 (0.4): IgPro20 (0.4 g/kg body weight): 20% liquid formulation (200 mg/mL) of human normal immunoglobulin for subcutaneous use administered weekly during the SC treatment period of the study according to the randomization.
- IgPro20 (0.2): IgPro20 (0.2 g/kg body weight): 20% liquid formulation (200 mg/mL) of human normal immunoglobulin for subcutaneous use administered weekly during the SC treatment period of the study according to the randomization.
Arm/Group | IgPro20 (0.4) | IgPro20 (0.2) | Placebo
Number analyzed (Participants) | 58 | 57 | 57
percentage of subjects | 32.8 | 38.6 | 63.2
Statistical Analysis 1: Comparison: IgPro20 (0.2) vs Placebo; Test type: Superiority; p = 0.007, Fisher Exact; Difference in Percent = -24.6, 95% CI 2-sided [-40.7 to -6.21]
Statistical Analysis 2: Comparison: IgPro20 (0.4) vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact; Difference in Percent = -30.4, 95% CI 2-sided [-46.0 to -12.2]

2. Secondary Outcome: Change in Inflammatory Neuropathy Cause and Treatment (INCAT) Scores During the SC Treatment Period
Description: The INCAT score is a 10-point scale that covers the functionality of legs and arms, and has been successfully used to measure treatment effects in various CIDP studies. Scores for arm disability range from 0 ("No upper limb problems") to 5 ("Inability to use either arm for any purposeful movement"), and scores for leg disability range from 0 ("Walking not affected") to 5 ("Restricted to wheelchair, unable to stand and walk a few steps with help"). The INCAT (total) score is the sum of these 2 scores and ranges from 0 to 10. For the "adjusted" INCAT score, changes in the function of the upper limbs from 0 (normal) to 1 (minor symptoms) or from 1 to 0 were not recorded as deterioration or improvement because these changes are not considered clinically significant.
Time Frame: Baseline and up to 25 weeks
Population: ITTS. Not all subjects from the ITTS were available for data collection for this outcome measure.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | IgPro20 (0.4) | IgPro20 (0.2) | Placebo
Number analyzed (Participants) | 57 | 56 | 57
units on a scale | 0 [-2 to 3] | 0 [-2 to 5] | 1 [-1 to 4]
Statistical Analysis 1: Comparison: IgPro20 (0.2) vs Placebo; Test type: Other; p = 0.005, Wilcoxon rank sum; Median Difference (Net) = 0, 95% CI 2-sided [-1 to 0]
Statistical Analysis 2: Comparison: IgPro20 (0.4) vs Placebo; Test type: Other; p < 0.001, Wilcoxon rank sum; Median Difference (Net) = -1, 95% CI 2-sided [-1 to 0]

3. Secondary Outcome: Median Change From Baseline in the Mean Grip Strength Scores of the Dominant Hand During the SC Treatment Period
Description: The hand-held Vigorimeter is a device that measures the strength of small muscles in the hand; ie, grip strength. Subjects squeezed a rubber bulb lying between the palm of the hand and the thumb and index fingers. The pressure was recorded via a rubber tube on a nanometer and expressed in kilopascal. At each assessment, the subjects squeezed 3 times with each hand. The mean grip strength median score of the dominant hand was determined.
Time Frame: Baseline and up to 25 weeks
Population: ITTS. Not all subjects from the ITTS were available for data collection for this outcome measure..
Measure: Median (Full Range); unit: Kilopascal (kPa)
Arm/Group | IgPro20 (0.4) | IgPro20 (0.2) | Placebo
Number analyzed (Participants) | 57 | 56 | 57
Kilopascal (kPa) | -2.7 [-80 to 55] | -0.6 [-80 to 55] | -6.6 [-51 to 22]
Statistical Analysis 1: Comparison: IgPro20 (0.2) vs Placebo; Test type: Other; p = 0.004, Wilcoxon rank sum; Median Difference (Net) = 7.6, 95% CI 2-sided [2 to 14]
Statistical Analysis 2: Comparison: IgPro20 (0.4) vs Placebo; Test type: Other; p = 0.014, Wilcoxon rank sum; Median Difference (Net) = 5.7, 95% CI 2-sided [0.7 to 11.7]

4. Secondary Outcome: Change in the Medical Research Council (MRC) Sum Scores During the SC Treatment Period
Description: An adapted version of the MRC sum score was used in the study. The MRC sum score is the sum of all 16 muscle scores, and ranges from 0 (paralysis) to 80 (normal strength).
Time Frame: Baseline and up to 25 weeks
Population: ITTS. Not all subjects from the ITTS were available for data collection for this outcome measure.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | IgPro20 (0.4) | IgPro20 (0.2) | Placebo
Number analyzed (Participants) | 57 | 56 | 57
units on a scale | 0 [-12 to 7] | 0 [-16 to 14] | -2 [-19 to 6]
Statistical Analysis 1: Comparison: IgPro20 (0.2) vs Placebo; Test type: Other; p = 0.003, Wilcoxon rank sum; Median Difference (Final Values) = 2, 95% CI 2-sided [1 to 4]
Statistical Analysis 2: Comparison: IgPro20 (0.4) vs Placebo; Test type: Other; p = 0.002, Wilcoxon rank sum; Median Difference (Final Values) = 2, 95% CI 2-sided [1 to 4]

5. Secondary Outcome: Change in Rasch-built Overall Disability Scale (R-ODS) Scores During the SC Treatment Period
Description: The R-ODS centile score captures activity and social participation in subjects with CIDP. The R-ODS centile score ranges from 0 (most severe activity and social participation limitations) to 100 (no activity and social participation limitations).
Time Frame: Baseline and up to 25 weeks
Population: ITTS. Not all subjects from the ITTS were available for data collection for this outcome measure.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | IgPro20 (0.4) | IgPro20 (0.2) | Placebo
Number analyzed (Participants) | 53 | 53 | 52
units on a scale | 0 [-49 to 17] | -2 [-41 to 100] | -3 [-43 to 13]
Statistical Analysis 1: Comparison: IgPro20 (0.2) vs Placebo; Test type: Other; p = 0.03, Wilcoxon rank sum; Median Difference (Net) = 3, 95% CI 2-sided [0 to 9]
Statistical Analysis 2: Comparison: IgPro20 (0.4) vs Placebo; Test type: Other; p < 0.001, Wilcoxon rank sum; Median Difference (Net) = 5, 95% CI 2-sided [2 to 9]

6. Secondary Outcome: Time to CIDP Relapse or Withdrawal Due to Any Other Reason During the SC Treatment Period
Time Frame: Up to 25 weeks
Population: ITTS
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | IgPro20 (0.4) | IgPro20 (0.2) | Placebo
Number analyzed (Participants) | 58 | 57 | 57
Days | NA [NA to NA] — Median times could not be calculated due to insufficient number of participants with events | NA [113.0 to NA] — Median times could not be calculated due to insufficient number of participants with events | 79.0 [57.0 to 125.0]

7. Secondary Outcome: Number of Adverse Events Per IgPro20 Infusion During the SC Treatment Period
Time Frame: Up to 28 weeks
Population: Safety Data Set (SDS): The SDS consists of all randomized subjects who received at least 1 dose of IgPro20 or placebo.
Measure: Number; unit: Adverse events/Infusion
Arm/Group | IgPro20 (0.4) | IgPro20 (0.2) | Placebo
Number analyzed (Participants) | 58 | 57 | 57
Adverse events/Infusion | 0.051 | 0.079 | 0.034

8. Secondary Outcome: Number of Subjects With Adverse Events During the SC Treatment Period
Time Frame: Up to 28 weeks
Population: SDS
Measure: Count of Participants; unit: Participants
Arm/Group | IgPro20 (0.4) | IgPro20 (0.2) | Placebo
Number analyzed (Participants) | 58 | 57 | 57
Participants | 30 | 33 | 21

9. Secondary Outcome: Percentage of Subjects With Adverse Events During the SC Treatment Period
Time Frame: Up to 28 weeks
Population: SDS
Measure: Number; unit: percentage of subjects
Arm/Group | IgPro20 (0.4) | IgPro20 (0.2) | Placebo
Number analyzed (Participants) | 58 | 57 | 57
percentage of subjects | 51.7 | 57.9 | 36.8

10. Secondary Outcome: Time to Improvement During IgPro10 Re-stabilization Therapy
Description: Improvement is defined as an INCAT score decrease by 1 point (except for the decrease from 1 to 0 in the upper limb score), R-ODS improvement by at least 4 points, Mean Grip strength improvement by at least 8 kPa in one hand, or MRC Sum score >=3.
Time Frame: Up to 13 weeks
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- IgPro10: Subjects who experienced CIDP deterioration during IgG Dependency received IVIG treatment with IgPro10 during IgPro10 Restabilization.
  IgPro10 as 1 loading dose of 2 g/kg bw, followed by 3 or 4 maintenance doses (depending on time needed for restabilization) of 1 g/kg bw every 3 weeks.
Arm/Group | IgPro10
Number analyzed (Participants) | 207
Days | 23 [22 to 23]

11. Secondary Outcome: Change in Mean Grip Strength During IgPro10 Re-stabilization Therapy
Description: as for outcome 3
Time Frame: Reference visit and up to 13 weeks
Population: PSDS. Not all subjects from the PSDS were available for data collection for this outcome measure.
Measure: Mean (Standard Deviation); unit: kPa
Groups:
- IgPro10: Subjects who experienced CIDP deterioration during IgG Dependency received IVIG treatment with IgPro10 during the IgPro10 Restabilization.
  IgPro10 as 1 loading dose of 2 g/kg bw, followed by 3 or 4 maintenance doses (depending on time needed for restabilization) of 1 g/kg bw every 3 weeks.
Arm/Group | IgPro10
Number analyzed (Participants) | 202
kPa | 11.27 (16.89)

12. Secondary Outcome: Change in MRC Sum Score During IgPro10 Re-stabilization Therapy
Description: as for outcome 4
Time Frame: Reference visit and up to 13 weeks
Population: PSDS. Not all subjects from the PSDS were available for data collection for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IgPro10
Number analyzed (Participants) | 203
units on a scale | 3.4 (4.9)

13. Secondary Outcome: Change in R-ODS During IgPro10 Re-stabilization Therapy
Description: as for outcome 5
Time Frame: Reference visit and up to 13 weeks
Population: PSDS. Not all subjects from the PSDS were available for data collection for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IgPro10
Number analyzed (Participants) | 166
units on a scale | 4.7 (14.14)

14. Secondary Outcome: Change in INCAT During IgPro10 Re-stabilization Therapy
Description: as for outcome 2
Time Frame: Reference visit and up to 13 weeks
Population: PSDS. Not all subjects from the PSDS were available for data collection for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IgPro10
Number analyzed (Participants) | 205
units on a scale | -1.1 (1.2)

15. Secondary Outcome: Number of Adverse Events Per IgPro10 Infusion During Re-stabilization Therapy
Time Frame: Up to 13 weeks
Population: PSDS
Measure: Number; unit: Adverse events/Infusion
Arm/Group | IgPro10
Number analyzed (Participants) | 207
Adverse events/Infusion | 0.175

16. Secondary Outcome: Number of Subjects With Adverse Events During IgPro10 Re-stabilization Therapy
Time Frame: Up to 13 weeks
Population: PSDS
Measure: Number; unit: participants
Arm/Group | IgPro10
Number analyzed (Participants) | 207
participants | 100

17. Secondary Outcome: Percent of Subjects With Adverse Events During IgPro10 Re-stabilization Therapy
Time Frame: Up to 13 weeks
Population: PSDS
Measure: Number; unit: percentage of subjects
Arm/Group | IgPro10
Number analyzed (Participants) | 207
percentage of subjects | 48.3

18. Secondary Outcome: Time to Improvement After CIDP Relapse During IgPro10 Rescue Therapy
Description: Improvement is defined as a decrease in INCAT score (except for the decrease from 1 to 0 in the upper limb score) back to or below the baseline score..The INCAT score is a 10-point scale that covers the functionality of legs and arms, and has been successfully used to measure treatment effects in various CIDP studies. Scores for arm disability range from 0 ("No upper limb problems") to 5 ("Inability to use either arm for any purposeful movement"), and scores for leg disability range from 0 ("Walking not affected") to 5 ("Restricted to wheelchair, unable to stand and walk a few steps with help"). The INCAT (total) score is the sum of these 2 scores and ranges from 0 to 10. For the "adjusted" INCAT score, changes in the function of the upper limbs from 0 (normal) to 1 (minor symptoms) or from 1 to 0 were not recorded as deterioration or improvement because these changes are not considered clinically significant.
Time Frame: Up to 13 weeks
Population: Rescue Medication Safety Data Set (RSDS): The RSDS consists of subjects of the SDS who received at least 1 dose of IgPro10 rescue medication.
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- IgPro10: Subjects who experienced CIDP relapse during the IgPro20 SC Period received IVIG treatment with IgPro10 during the IgPro10 Rescue.
  IgPro10 as 1 loading dose of 2 g/kg bw, followed by 3 or 4 maintenance doses of 1 g/kg bw every 3 weeks.
Arm/Group | IgPro10
Number analyzed (Participants) | 60
Days | 23 [22 to 49]

19. Secondary Outcome: Number of Adverse Events Per IgPro10 Infusion During Rescue Therapy
Time Frame: Up to 13 weeks
Population: RSDS
Measure: Number; unit: Adverse events/Infusion
Arm/Group | IgPro10
Number analyzed (Participants) | 60
Adverse events/Infusion | 0.142

20. Secondary Outcome: Number of Subjects With Adverse Events During IgPro10 Rescue Therapy
Time Frame: Up to 13 weeks
Population: RSDS
Measure: Number; unit: participants
Arm/Group | IgPro10
Number analyzed (Participants) | 60
participants | 17

21. Secondary Outcome: Percent of Subjects With Adverse Events During IgPro10 Rescue Therapy
Time Frame: Up to 13 weeks
Population: RSDS
Measure: Number; unit: percentage of subjects
Arm/Group | IgPro10
Number analyzed (Participants) | 60
percentage of subjects | 28.3

22. Secondary Outcome: Change in Mean Grip Strength During IgPro10 Rescue Therapy
Description: as for outcome 3
Time Frame: Before first rescue IgPro10 infusion and up to 13 weeks
Population: RSDS. Not all subjects from the RSDS were available for data collection for this outcome measure.
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | IgPro10
Number analyzed (Participants) | 35
kPa | 16.3 (17.58)

23. Secondary Outcome: Change in MRC Sum Score During IgPro10 Rescue Therapy
Description: as for outcome 4
Time Frame: Before first rescue IgPro10 infusion and up to 13 weeks
Population: RSDS. Not all subjects from the RSDS were available for data collection for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IgPro10
Number analyzed (Participants) | 35
units on a scale | 6.8 (5.28)

24. Secondary Outcome: Change in R-ODS During IgPro10 Rescue Therapy
Description: as for outcome 5
Time Frame: Before first rescue IgPro10 infusion and up to 13 weeks
Population: RSDS. Not all subjects from the RSDS were available for data collection for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IgPro10
Number analyzed (Participants) | 29
units on a scale | 14.0 (14.69)

25. Secondary Outcome: Change in INCAT During IgPro10 Rescue Therapy
Description: as for outcome 2
Time Frame: Before first rescue IgPro10 infusion and up to 13 weeks
Population: RSDS. Not all subjects from the RSDS were available for data collection for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IgPro10
Number analyzed (Participants) | 45
units on a scale | -1.3 (1.31)

ADVERSE EVENTS:
Time Frame: 4.5 years
Groups:
- IgPro10 Restabilization: IgPro10: 10% Immunoglobulin G (IgG) liquid formulation of human normal immunoglobulin (Privigen®) administered intravenously during restabilization.
  IgPro10 as 1 loading dose of 2 g/kg bw, followed by 3 or 4 maintenance doses (depending on time needed for restabilization) of 1 g/kg bw every 3 weeks.
- IgPro20 (0.4): IgPro20 (0.4 g/kg body weight): 20% liquid formulation (200 mg/mL) of human normal immunoglobulin for subcutaneous use administered weekly.
- IgPro20 (0.2): IgPro20 (0.2 g/kg body weight): 20% liquid formulation (200 mg/mL) of human normal immunoglobulin for subcutaneous use administered weekly.
- Placebo: Placebo: 2% human albumin administered by weekly SC infusions during the IgPro20 SC treatment period of the study.
- IgPro10 Rescue: IgPro10: 10% Immunoglobulin G (IgG) liquid formulation of human normal immunoglobulin (Privigen®) administered intravenously during rescue.
  IgPro10 as 1 loading dose of 2 g/kg bw, followed by 3 or 4 maintenance doses of 1 g/kg bw every 3 weeks.
Arm/Group | IgPro10 Restabilization | IgPro20 (0.4) | IgPro20 (0.2) | Placebo | IgPro10 Rescue
All-Cause Mortality (participants affected / at risk) | 0/207 | 0/58 | 0/57 | 0/57 | 0/60
Serious Adverse Events (participants affected / at risk) | 11/207 | 2/58 | 3/57 | 1/57 | 2/60
Other Adverse Events (participants affected / at risk) | 50/207 | 20/58 | 22/57 | 15/57 | 7/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IgPro10 Restabilization (N=207) | IgPro20 (0.4) (N=58) | IgPro20 (0.2) (N=57) | Placebo (N=57) | IgPro10 Rescue (N=60)
Blood pressure diastolic increased (Investigations) | 1 | 0 | 0 | 0 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Choleithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IgPro10 Restabilization (N=207) | IgPro20 (0.4) (N=58) | IgPro20 (0.2) (N=57) | Placebo (N=57) | IgPro10 Rescue (N=60)
Fall (Injury, poisoning and procedural complications) | 5 (5) | 1 (1) | 3 (8) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 34 (53) | 4 (4) | 4 (5) | 2 (2) | 4 (6)
Fatigue (General disorders) | 5 (11) | 0 (0) | 5 (5) | 1 (1) | 0 (0)
Infusion site erythema (General disorders) | 0 (0) | 10 (28) | 5 (11) | 0 (0) | 0 (0)
Infusion site swelling (General disorders) | 0 (0) | 6 (8) | 5 (8) | 2 (2) | 0 (0)
Infusion site induration (General disorders) | 0 (0) | 3 (3) | 2 (10) | 1 (1) | 0 (0)
Infusion site pain (General disorders) | 0 (0) | 2 (2) | 3 (15) | 2 (2) | 0 (0)
Infusion site warmth (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 10 (12) | 1 (1) | 0 (0) | 2 (2) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1) | 3 (4) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 12 (12) | 2 (2) | 4 (6) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2) | 3 (3) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
CSL agreements may vary with individual investigators; however, CSL will not prohibit any investigator from publishing. CSL supports the publication of results from all centers of a multi-center trial and requests that reports based on single-site data not precede the primary publication of the entire clinical trial.